CLINICAL TRIAL: NCT06334445
Title: CARDIOCARE Prospective Clinical Study An Interdisciplinary Approach for the Management of the Elderly Multimorbid Patient With Breast Cancer Therapy Induced Cardiac Toxicity
Brief Title: CARDIOCARE Prospective Clinical Study
Acronym: CARDIOCARE
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1874
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Wearables/sensors and ePsycHeart App
  Interventions: Behavioral: Control group
- Intervention group: Wearables/sensors and ePsycHeart App and eHealtHeart
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Control group — Wearables/sensors and ePsycHeart App
  Groups: Control group
Behavioral: Intervention group — Wearables/sensors and ePsycHeart App and eHealtHeart
  Groups: Intervention group

SUMMARY:
This is a prospective observational study to refine and validate risk stratification algorithms aimed at identifying elderly patients at higher risk of developing cardiotoxicity (us-ing risk factors and potential blood and stool biomarkers) and at assessing whether integrated patient-oriented behavioral and psychological interventions can mitigate, prevent or delay the onset of cardiotoxicity from chemotherapy.

DETAILED DESCRIPTION:
This is a prospective observational study for women with diagnosis of Breast Cancer (BC) who will undergo neoadjuvant and/or adjuvant treatment:

1. Women ≥ 60 years with a diagnosis of HER2-positive early/locoregional breast cancer with anti-HER2 therapy (trastuzumab or trastuzumab and pertuzumab)
2. Women ≥ 60 years with a diagnosis of early/locoregional breast cancer who will un-dergo neoadjuvant and/or adjuvant treatment with regimens including anthracy-clines and/or taxanes
3. Women ≥60 years with a diagnosis of early/locoregional breast cancer who will un-dergo neoadjuvant and/or adjuvant treatment with endocrine therapies +/- CDK 4/6 inhibitors
4. Women ≥ 60 years with HER2-positive metastatic breast cancer who will undergo first-line therapy with anti-HER2 therapy (trastuzumab or trastuzumab and per-tuzumab +/- chemotherapy).

The study primary objective is to evaluate the onset of cardiotoxicity, where: subclinical car-diotoxicity is defined as preserved Left Ventricular Ejection Fraction (LVEF).

All patients will receive, in addition to standard of care, supportive care. Patients in the control and in the intervention group will receive wearable and will be invited to complete the mobile ePsycHeart evaluation. ePsycHeart will assess patients' intrinsic capacity indicators that may be associated with including

1. psycho cognitive states (psychological and emotional states, QoL, cognitive function and memory, perceptions of aging, environmental and social factors),
2. mobility and locomotion (distance, balance, gait speed), and
3. vitality (exercise, electrocardiogram (ECG), Heart Rate Variability (HRV), grip strength, nutritional/energy state, sleep, fatigue), will be performed by means of sensors, wearables, electronic devices and validated patient reported outcome- and experience measures.

In addition, patients in the intervention group will receive the eHealtHeart: Behavioral and psychological interventions will be delivered to the intervention arm via the eHealtHeart mobile application to mitigate potential risk factors associated with cardiotoxicity and deterioration of QoL. eHealtHeart interventions will target patients and care givers aiming at improving patients' intrinsic capacity including psychological inter-ventions (e.g. emotional, dispositional states, biofeedback self-regulation, best possible self), cognitive stim-ulation (e.g. cognitive restructuring plus card games to improve memory and executive functions), sensory screening, physical activity and performance exercises, vision and hearing suggestions, dietary guidance on nutrition, guidance to improve management of urinary inconti-nence (e.g. alerts, self-monitoring) and falls together with providing education and support to caregivers. At month 6 the patient will have to return the wearables used for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 60 years with a diagnosis of early/locoregional breast cancer who will undergo neoadju-vant and/or adjuvant treatment with regimens including anthracyclines and/or taxanes.
2. Women ≥ 60 years with a diagnosis of HER2-positive locoregional breast cancer who will undergo neoadjuvant and/or adjuvant treatment with anti-HER2 therapy (trastuzumab or trastuzumab and pertuzumab).
3. Women ≥ 60 years with a diagnosis of early/locoregional breast cancer who will undergo neoadju-vant and/or adjuvant treatment with endocrine therapies +/- CDK 4/6 inhibitors.
4. Women ≥ 60 years with HER2-positive metastatic breast cancer who will undergo first-line therapy with anti-HER2 therapy (trastuzumab or trastuzumab and pertuzumab +/- chemotherapy).
5. Women with age ≥ 60 years before starting the aforementioned treatment for breast cancer.
6. Women eligible ≥ 60 years who will undergo first-line therapy in the metastatic setting with any type of treatment (chemotherapy, immunotherapy, biological agents).
7. Willingness and ability to comply with scheduled visits, laboratory tests, and other trial procedures
8. Written informed consent.
9. Participant affiliated to a social security system.
10. Life expectancy of at least 12 months.

Exclusion Criteria:

1. Age < 60 years.
2. Diagnosed severe psychiatric or neurological disorders that might impair the ability to give informed consent.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective clinical study will enroll a total of 750 breast cancer patients over 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 736 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the onset of cardiotoxicity | 12 months
  Subclinical cardiotoxicity is defined as preserved Left Ventricular Ejection Fraction (LVEF) with >15% reduction in Global Longitudinal Strain (GLS) relative to baseline and/or new rise in cardiac Troponin I or Natriuretic peptides levels in plasma.
  Clinical cardiotoxicity is defined as the reduction of LVEF by ≥ 10% from baseline to a value below 50%, incurred at any timepoint during study Follow Up (FU)

SECONDARY OUTCOMES:
Intra-patient assessment of major adverse cardiac events (MACEs) | 12 months
  1. Angina pectoris;
  2. Acute myocardial infarction;
  3. Major ventricular arrhythmias;
  4. Pacemaker implantation;
  5. Acute heart failure (New York Heart Association (NYHA) class 4);
  6. Acute ischemic brain disease with neurological persistence evidence;
  7. Severe hypertension requiring treatment with Angiotensin-converting enzyme (ACE) and or beta blockers.
Intra-patient assessment of plasma Troponin I | 12 months
  Intra-patient assessment of plasma Troponin I during follow up and association/agreement with LVEF
Intra-patient assessment of plasma Brain natriuretic peptide (BNP) elevation | 12 months
  Intra-patient assessment of plasma Brain natriuretic peptide (BNP) elevation
Percentage in the two arm of hospital admission | 12 months
  Hospital admissions from cardiovascular causes or falls in order to evaluate the percentage in the two arms
Number of Cardiovascular death in the two arms | 12 months
  Number of Cardiovascular death in the two arms
Number of Non-cardiovascular death in the two arms | 12 months
  Number of Non-cardiovascular death in the two arms
Evaluation of Health Related Quality of Life in the two arms | 12 months
  Evaluation of Health Related Quality of Life in the two arms assessed by EORTC QLQ-BR23, validated breast cancer Patient Re-ported Outcome Measure (PROM)
Cost-effectiveness of provided healthcare pathways determined by costs combined with quality-adjusted life-years (QALYs) in the two arms | 12 months
  Cost-effectiveness of provided healthcare pathways determined by costs combined with quality-ad-justed life-years (QALYs). Costs will consider healthcare provided, numbers of admission and days spent in hospital and patient costs for out-of-pocket expenses associated with their condition (i.e., travel expenses (of both patient and caregiver), over-the-counter medicines and supplements, com-plementary therapies not supported by Healthcare system, home help, and time away from work).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Sacco GGA, Mazzocco K, Constantinidou A, Papakonstantinou A, Mauri D, Kalliatakis G, Tsiknakis M, Ribnikar D, Tsekoura D, Aidarinis V, Keramida K, Oikonomopoulos P, Antoniades A, Brown C, Rizzi F, Bucur A, Pacella E, Karanasiou G, Cardinale D, Cipolla C, Munzone E, Fotiadis D, Curigliano G, Pravettoni G. An Interdisciplinary Ecosystem for the Prevention of Cardiotoxicity in Older Patients With Breast Cancer: Protocol for a Prospective and Multicentric Study. JMIR Res Protoc. 2025 Aug 14;14:e63455. doi: 10.2196/63455. PMID 40810441